CLINICAL TRIAL: NCT00490893
Title: Effects of Insulin Detemir Versus Regular Insulin (Actrapid) on Hormonal Counterregulation, Cognitive Function and Symptom Perception During Hypoglycemia
Brief Title: Hypoglycemia Counterregulation and Symptom Perception With Insulin Detemir
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 2005-003940-79
Record Dates: First submitted 2007-06-22; First posted 2007-06-25 (Estimated); Last update posted 2007-06-25 (Estimated); Status verified 2007-06

CONDITIONS: Diabetes Mellitus; Hypoglycemia
Keywords: counterregulation; hypoglycemia unawareness; insulin therapy
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Detemir

SUMMARY:
Hypoglycemia and unawareness of hypoglycemia are major problems of insulin therapy in patients with diabetes mellitus. The long acting insulin analogue Detemir has structural and physicochemical properties which differ from human insulin. The aim of the present study is to test whether this leads to altered hormone and symptom response during hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects male or female
* Age 18-50 years
* Female subjects save contraception
* Ability to take part in the study
* Signed consent

Exclusion Criteria:

* Chronic disease
* Acute disease during 4 weeks prior to the study
* Pregnancy
* Drug treatment other than hormonal contraception

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-03; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Hormone response to hypoglycemia (Glucagon)
Hormone response to hypoglycemia (glucagon) Symptom response to hypoglycemia

SECONDARY OUTCOMES:
Hormone response to glucagon (epinephrine, growth hormne, cortisol)
Hormone response (epinephrine, growth hormone, cortisol) to hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Fritsche, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University of Tübingen, Medical Department, Tübingen, Germany